CLINICAL TRIAL: NCT02385344
Title: Registry for Quality Assessment With Ultrasound Imaging and TTFM in Cardiac Bypass Surgery
Acronym: REQUEST
Status: Completed | Type: Observational
Sponsor: Medistim ASA (Industry)
Responsible Party: Sponsor
Other Study IDs: 1501
Record Dates: First submitted 2015-02-17; First posted 2015-03-11 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Medistim device — This registry is intended to document surgical findings, procedural changes, and adverse events occurring prior to discharge

SUMMARY:
The purpose of the registry is to collect information regarding the number and type of coronary artery bypass (CAB) surgical procedure changes that are made based on intraoperative guidance information using transit time flow measurements (TTFM) and ultrasound image capabilities provided with the Medistim device.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been scheduled for coronary bypass surgery
* Subject understands the nature of the procedure and has signed the subject informed consent prior to the procedure
* Subject has been diagnosed with 2-3 vessel disease

Exclusion Criteria:

* Subject is scheduled for other surgical procedures during the bypass surgery (valve replacement/repair, carotid endarterectomy, etc.)
* Subject is known to be suffering from any psychological, developmental, physical, or emotional disorder that the investigator feels would interfere with surgery or follow-up testing
* Subject is undergoing an emergency cardiac bypass surgery
* Subject has history or presence of muscle disease (i.e. myopathy, myalgia, myasthenia, rhabdomyolysis) with or without concomitant CK-elevation > 5 ULN that cannot be ascribed to any other medical condition (e.g. myocardial infarction)
* Subject has any condition that the investigator believes should exclude him/her from this registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject has been scheduled for coronary bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in planned surgical procedure | Day 1 (During Surgery)
  Identify how often epiaortic scanning With the Medistim Device, leads to a change in the planned surgical procedure and to identify the reason and the procedure change
Procedure adaptions | Day 1 (During surgery)
  Identify the procedure adaptions made by a surgeon when TTFM and/or Medistim ultrasound imaging identify suboptimal graft function

SECONDARY OUTCOMES:
Record number of revisions | Day 1 (During surgery)
  Record how many Cardiac bypass patients experience intraoperative graft revision, the type of revision, and the key identifier motivating the revision
Record number of events | Day 1-14 (During hospitalization)
  Record post-surgical major adverse cardiac and cerebral events (MACCE) of all bypass procedure patients entered into the registry and occuring prior to discharge
Incidence rate | 2 years (Throughout the study)
  To determine the incidence rate of Serious Adverse Events (SAE) and/or Unanticipated Adverse Events (UAE) throughout the registry

CONTACTS AND LOCATIONS:
Overall Officials: Anne Waaler, MSc Pharm, Study Director — Medistim ASA
Locations (7):
- United States (2):
  - Veterans Affairs Medical Center, Washington DC, Maryland
  - Mount Sinai Beth Israel, New York, New York
- University of Calgary, Calgary, Alberta, Canada
- University of Duisburg-Essen, Dept. of Cardiothoracic Surgery, Essen, Germany
- Clinica Cardiochirurgica, Chieti, Italy
- Erasmus University Medical Center, Rotterdam, Netherlands
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Leviner DB, von Mucke Similon M, Rosati CM, Amabile A, Thuijs DJFM, Giammarco GD, Wendt D, Trachiotis GD, Kieser TM, Kappetein AP, Head SJ, Taggart DP, Puskas JD. Transit time flow measurement of coronary bypass grafts before and after protamine administration. J Cardiothorac Surg. 2021 Jul 9;16(1):195. doi: 10.1186/s13019-021-01575-y. PMID 34243799
- [Derived] Rosenfeld ES, Trachiotis GD, Napolitano MA, Sparks AD, Wendt D, Kieser TM, Puskas JD, DiGiammarco G, Taggart DP. Intraoperative transit-time flow measurement and high-frequency ultrasound in coronary artery bypass grafting: impact in off versus on-pump, arterial versus venous grafting and cardiac territory grafted. Eur J Cardiothorac Surg. 2021 Dec 27;61(1):204-213. doi: 10.1093/ejcts/ezab239. PMID 34166508
- [Derived] Rosenfeld ES, Trachiotis GD, Sparks AD, Napolitano MA, Lee KB, Wendt D, Kieser TM, Puskas JD, DiGiammarco G, Taggart DP. Intraoperative surgical strategy changes in patients with chronic and end-stage renal disease undergoing coronary artery bypass grafting. Eur J Cardiothorac Surg. 2021 Jun 14;59(6):1210-1217. doi: 10.1093/ejcts/ezab104. PMID 33675642